CLINICAL TRIAL: NCT06237075
Title: Combining Functional Magnetic Resonance Imaging and Transcranial Direct Current Stimulation to Investigate Pain-related Brain Networks in Patients With Neuropathic Pain
Brief Title: Combining fMRI and tDCS in Neuropathic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202012283RINA
Record Dates: First submitted 2024-01-15; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Patients with neuropathic pain versus healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS stimulation (Experimental): 2-milliamp stimulation for 5~15 min
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — 2-milliamp stimulation for 5~15 min

SUMMARY:
The proposed project aims to explore possible neuromodulatory effects of transcranial direct current stimulation (tDCS) on neuropathic pain caused by peripheral neuropathy. tDCS will be performed through an MRI-compatible stimulation setting during functional magnetic resonance imaging (fMRI) scanning. The stimulation target of tDCS will be the primary motor cortex (M1) and the dorsolateral prefrontal cortex (DLPFC). We expect that results from the current project will advance the understanding of neuromodulatory mechanisms of tDCS and facilitate the development of treatment strategies for patients with neuropathic pain.

DETAILED DESCRIPTION:
Neuropathic pain is the most excruciating symptom in peripheral neuropathy such as diabetic or chemotherapy-induced neuropathy. Management of neuropathic pain is a challenging clinical problem because only less than 50% patients are responsive to pharmacological treatment. Neuropathic pain is naturally considered as a direct consequence of peripheral nerve injury that induces hypersensitivity or ectopic activities in nociceptive nerve terminals. Nevertheless, maladaptive changes in the pain-related networks of the brain also play a crucial role in the generation, amplification, and drug-resistance of neuropathic pain. The proposed project aims to explore possible neuromodulatory effects of transcranial direct current stimulation (tDCS) on neuropathic pain caused by peripheral neuropathy. tDCS is a non-invasive stimulation technique that delivers a low-intensity current into the brain to modulate the synaptic plasticity of cortical neurons. To investigate the instantaneous effects of tDCS, tDCS will be performed through an MRI-compatible stimulation setting during functional magnetic resonance imaging (fMRI) scanning. The stimulation target of tDCS will be the primary motor cortex (M1) and the dorsolateral prefrontal cortex (DLPFC). This simultaneous tDCS-fMRI approach will enable us to (1) identify the neural substrates of neuropathic pain that could be modulated by neurostimulation, (2) to characterize the spatial patterns of functional hemodynamic brain responses following tDCS, and (3) to assess changes in cortical excitability and neuroplasticity associated with pain perception after non-invasive brain stimulation. We expect that results from the current project will advance the understanding of neuromodulatory mechanisms of tDCS and facilitate the development of treatment strategies for patients with neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 20 or older and 90 or younger. 2. Ability to give informed consent 3. Neuropathic pain and/or nonpainful sensory symptoms resulted from I or II I. Peripheral neuropathy confirmed by clinical symptoms nerve conduction study, autonomic function test, quantitative sensory test, or skin biopsy.

II. Stroke involving somatosensory pathway confirmed by neuroimage 4. Agree not to take caffeine, alcohol, tea and drugs with significant nervous system effects for 48 hours before each study session.

Exclusion Criteria:

* 1. Presence of sever systemic diseases, including severe ischemic heart disease or congestive heart failure (left ventricular ejection fraction < 30%), severe lung diseases with dyspnea, severe generalized edema, and systemic infection 2. Presence of major neurological disorders, including brain tumor, head trauma and infection or inflammation of nervous system.

  3. Presence of major depression or any major mental disorders 4. Presence of a cardiac pacemaker, brain stimulator, aneurysm clips or metal implants in the head, unless these devices are certified to be MRI-compatible 5. Pregnancy 6. Claustrophobia or any other contraindications to MRI 7. Inability to give informed consent.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2030-09-11 (Estimated); Study Completion 2030-09-11 (Estimated)

PRIMARY OUTCOMES:
Brain functional connectivity changes | 5 days after stimulation
  changes in brain functional connectivity after tDCS, assessed using functional MRI

SECONDARY OUTCOMES:
Intensity of neuropathic pain | 5 days after stimulation
  reduction of neuropathic pain assessed using visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No